CLINICAL TRIAL: NCT00005886
Title: A Phase IB Randomized Study of an Antiestrogen in Women With Newly Diagnosed Breast Cancer
Brief Title: Tamoxifen Compared With LY353381 in Treating Women With Newly Diagnosed Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000067956; KUMC-7813-99; KUMC-HSC-7419-98; NCI-P00-0158
Record Dates: First submitted 2000-06-02; First posted 2003-08-29 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; ductal breast carcinoma in situ; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Tamoxifen

INTERVENTIONS:
Drug: arzoxifene hydrochloride
Drug: tamoxifen citrate

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using tamoxifen or LY353381 may fight breast cancer by blocking the use of estrogen.

PURPOSE: This randomized phase I trial is studying how well tamoxifen works on the biomarkers of the tumor tissue, compared with LY353381, in treating women with newly diagnosed breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether LY353381 hydrochloride or tamoxifen administered in the interval between biopsy and re-excision alters the expression of tissue biomarkers relative to placebo controls in postmenopausal women with newly diagnosed breast cancer.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study.

* Phase I: Patients are randomized to receive either oral LY353381 hydrochloride or oral placebo daily.

Upon completion of phase I, all treatment centers begin phase II of the study.

* Phase II: Patients are randomized to receive either oral tamoxifen or oral placebo daily.

Treatment in both phases continues for 2-6 weeks (until scheduled lumpectomy or mastectomy) in the absence of disease progression or unacceptable toxicity.

Patients are followed at 1 and 2 weeks after surgery.

PROJECTED ACCRUAL: A minimum of 120 patients (60 per treatment phase) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed noninvasive or small invasive breast cancer

  * Low or intermediate grade (ductal carcinoma in situ, T1, or T2) OR
  * Estrogen and/or progesterone receptor positive
  * Largest mass no greater than 5 cm
  * Clustered microcalcifications as only abnormality allowed with no upper size limit
  * If no distinction between mass and microcalcifications, size as 1 lesion
* Lumpectomy or mastectomy must be planned for 2-6 weeks from start of study
* No evidence of metastases from any malignancy
* Hormone receptor status:

  * Estrogen and progesterone receptor positive (unless low or intermediate grade tumor)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Postmenopausal by one of the following:

  * Prior oophorectomy
  * Over age 50 with prior hysterectomy, ovaries remaining
  * Uterus and ovaries intact and no menstrual period for more than 3 months

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 10 g/dL
* Absolute granulocyte count greater than 1,000/mm^3

Hepatic:

* Albumin greater than 3 g/dL
* Bilirubin less than 1.5 mg/dL
* AST less than 100 U/L
* Alkaline phosphatase less than 200 U/L

Renal:

* Creatinine less than 1.5 mg/dL

Cardiovascular:

* No history of deep vein thrombosis

Pulmonary:

* No prior pulmonary embolus

Other:

* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 1 year since prior chemotherapy

Endocrine therapy:

* At least 1 year since prior aromatase inhibitors, antiestrogens, or LH agonists/antagonists
* No concurrent hormone replacement therapy or oral contraceptives (from time of randomization)

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Other:

* No concurrent treatment for other malignancy

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-07; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol J. Fabian, MD, Study Chair — University of Kansas
Locations (9):
- United States (9):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Comprehensive Cancer Centers of the Desert, Palm Springs, California
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - U.S. Oncology Research Inc., Dallas, Texas

REFERENCES:
- [Background] Fabian CJ, Kimler BF, Anderson J, Tawfik OW, Mayo MS, Burak WE Jr, O'Shaughnessy JA, Albain KS, Hyams DM, Budd GT, Ganz PA, Sauter ER, Beenken SW, Grizzle WE, Fruehauf JP, Arneson DW, Bacus JW, Lagios MD, Johnson KA, Browne D. Breast cancer chemoprevention phase I evaluation of biomarker modulation by arzoxifene, a third generation selective estrogen receptor modulator. Clin Cancer Res. 2004 Aug 15;10(16):5403-17. doi: 10.1158/1078-0432.CCR-04-0171. PMID 15328178